CLINICAL TRIAL: NCT07079254
Title: Surgical Outcome After Displaced Bucket-handle Meniscal Lesions - Repair Versus Partial Meniscectomy: A 10-year Observational Study
Brief Title: Surgical Outcome After Displaced Bucket-handle Meniscal Lesions - Repair Versus Partial Meniscectomy
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-00059-01
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Meniscus Rupture; Meniscus Injury; Osteoarthritis of Knee
Keywords: Meniscus; Re-operation; Bucket-handle; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Meniscus suture — The meniscus bucket-handle injury will either be treated with meniscus suture or partial meniscectomy
Procedure: Partial meniscectomy — The meniscus bucket-handle injury wil be treated with either meniscus suture or partial meniscectomy

SUMMARY:
The menisci of the knee joint are structures composed of cartilage and connective tissue, whose primary functions are to stabilize the joint and distribute weight across joint surfaces. In doing so, it helps protect the joint from osteoarthritis - a form of joint failure commonly referred to as "joint wear". Meniscal surgeries are among the most common orthopaedic procedures performed both in Sweden and globally. Historically, damaged menisci were treated by removing the injured part. However, this approach is linked to early-onset osteoarthritis. Osteoarthritis affects approximately one-third of individuals over the age of 45 and ranks among the ten most common diagnoses in Europe based on years lived with disability. The knee is the most frequently affected joint, and the importance of the menisci in preserving knee function has become increasingly recognized.

In recent years, advances in surgical techniques have led to a shift towards meniscus-preserving procedures. A typical injury is the displaced meniscus, in which a large portion of the meniscus becomes detached from the joint capsule and wedges itself inside the joint, causing mechanical locking and preventing full extension. A displaced meniscus often loses its blood supply and suffers mechanical damage from being compressed between the joint surfaces. To preserve the meniscus and prevent irreversible damage, early surgical intervention is required. If the injury is too old or the tissue too damaged, the injured part of the meniscus must be removed, which significantly increases the risk of developing early knee osteoarthritis.

It remains unclear how soon surgery must be performed to successfully preserve the meniscus, and this likely depends on various other factors, including patient age, presence of additional joint injuries, and surgical technique. There is currently no reliable data on the proportion of displaced menisci that heal after meniscus-preserving surgery. However, studies suggest that 20-30% of repaired menisci require reoperation due to failed healing.

Given that displaced menisci are considered surgical emergencies, they pose a significant burden on healthcare systems already strained by limited access to urgent surgery. Meanwhile, ongoing development of surgical techniques raise ethical and logistical questions for health providers - especially as the scientific evidence for the benefits of some advanced treatments remains inconclusive.

Therefore, more research is needed to guide the optimal management of displaced bucket-handle lesions across a diverse patient population, taking into account age, activity level, and concurrent injuries. A key priority is to identify predictors of healing potential, particularly the time window during which surgical repair remains a viable option. With better knowledge, more menisci could potentially be preserved - reducing both the number of unnecessary re-operations and the long-term incidence of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* 15 years or above.
* Displaced longitudinal bucket-handle tear including the posterior horn on MRI and a knee extension deficit.

Exclusion Criteria:

* Patient younger than 15 years.
* Insufficient knowledge of the Swedish language.
* Per-operative findings including a bucket-handle rupture in combination with a complete radial rupture

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who present to the emergency department or the orthopaedic outpatient clinics at our hospitals with a knee extension deficit after trauma, with a clinically suspected bucket-handle meniscus rupture, are referred to a magnetic resonance imaging (MRI) within a week. Patients with a bucket-handle tear on the MRI, and no younger than 15 years, will be invited to participate in the study. Recruitment takes place at the outpatient clinic at the orthopaedic department at Skåne University Hospital in Malmö and the orthopaedic department at Hässleholm hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-10-07 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2045-12 (Estimated)

PRIMARY OUTCOMES:
Re-operation | 2-10 years
  Re-operation for meniscus injury/lesion

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | From 6 months to 10 years
  Patient reported outcome measure in the form of Knee Injury and Outcome Score (KOOS). A total score, called KOOS4, without the ADL scale, will be calculated. The scale ranges from 0 (worst) to 100 (best).
Osteoarthritis in the knee | 10 years
  Radiological osteoarthritis

CONTACTS AND LOCATIONS:
Overall Officials: Ola Svejme, MD, PhD, Principal Investigator — Lund University, Department of Orthopaedics, Clinical Sciences, Malmö, Sweden
Locations (2):
- Sweden (2):
  - Region Skåne, Orthopaedic department Kristianstad/Hässleholm, Hässleholm, Skåne County
  - Region Skåne, Skåne University Hospital, Malmo, Skåne County

IPD SHARING:
Plan to Share IPD: No
Contains sensitive data such as social security number and surgery references, etc